CLINICAL TRIAL: NCT03904225
Title: Efficacy and Safety Evaluation of Tegio Consolidation Therapy in the Treatment of Nasopharyngeal Carcinoma With High Risk of Metastasis: a Phase II Study
Brief Title: Tegio Consolidation Therapy for NPC Patients With High Risk of Metastasis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NPC 2018 Tegio
Record Dates: First submitted 2019-01-01; First posted 2019-04-05 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-04

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: adjuvant chemotherapy; Tegio
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — tegafur-gimeracil-oteracil

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tegio (Experimental): Tegio 60mg bid d1-28 q6wks was administered until disease progression, unacceptable toxicity,or over 12monthes within 3monthes after curative chemoradiation
  Interventions: Drug: Tegafur-Gimeracil-Oteracil
- control (No Intervention): patients was oberved

INTERVENTIONS:
Drug: Tegafur-Gimeracil-Oteracil — oral administration for 12 months
  Arms: tegio

SUMMARY:
oral administration of Tegio capsules for 12 months for NPC patients with high risk of metastasis (AJCC stage T3-4N2M0 or T1-4N3M0) was tested trying to reduce distant metastasis，safety was also evaluated.

DETAILED DESCRIPTION:
In this study, NPC patients (stage T3-4N2M0 or T1-4N3M0) who finished the curative chemoradiation will be randomized to the observation group and treatment group (60 mg bid, p.o.，d1-28，q6wks; continued until disease progression, unacceptable toxicity, or over 1 year). The primary endpoint is distant failure-free survival (D-FFS), Secondary end points include overall survival (OS), locoregional failure-free survival (LR-FFS), progression-free survival (PFS) and toxic effects,. All efficacy analyses are conducted in the intention-to-treat population, and the safety population include only patients who receive their randomly assigned treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 ys
2. Performance status of Eastern Cooperative Oncology Group (ECOG) grade 0 -2
3. Tumor staged as 8th American Joint Committee on Cance (AJCC) T3-4N2M0 or T1-4N3M0 with histologically confirmed
4. Within 12weeks after completion of the curative radiotherapy treatment
5. disease was controlled after radiotherapy
6. with adequate hematologic (neutrophil count > 1.5×10^9/L, hemoglobin > 90g/L and platelet count > 100×10^9/L), hepatic (alanine aminotransferase, aspartate aminotransferase ≤ 1.5×ULN, bilirubin ≤ 1.5×ULN, alkaline phosphatase < 2.5×ULN) and renal function (creatinine clearance > 50 ml/min)
7. Patients must be informed and written informed consent was finished.

Exclusion Criteria:

1. allergic to Tegio.
2. Illness may interfere with oral medication, including dysphagia, chronic diarrhea, or ileus
3. Prior malignancy except treated basal cell or in situ cervical cancer.
4. Pregnancy or lactation (consider pregnancy test in women of child-bearing age and emphasize effective contraception during the treatment period).
5. severe comorbidities may bring unacceptable risk or affect the compliance of the trial, including but not limited to unstable cardiac disease requiring treatment, renal disease, chronic hepatitis, diabetes with poor control (fasting plasma glucose > 1.5×ULN), and emotional disturbance.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2018-12-14 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
distant metastsis-free survival (DMFS) | From date of randomization until the date of first documented distant disease failure, assessed up to 36 months
  distant metastsis-free survival

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China